CLINICAL TRIAL: NCT06149377
Title: Application of a Predictive Model on Sentinel Lymph Node Biopsy in Initially Lymph Node-positive, HER2-positive Breast Cancer After Neoadjuvant Systemic Therapy: a Multicenter Retrospective Study
Brief Title: Impact of a Predictive Model on Sentinel Lymph Node Biopsy in Initially Lymph Node-positive, HER2-positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Chuan Wang, Head of department of breast surgery, Fujian Medical University Union Hospital
Other Study IDs: NSFFP-2023Y0020
Record Dates: First submitted 2023-11-04; First posted 2023-11-29 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort: Patients (n=386) who accepted neoadjuvant systemic therapy followed surgery were from fujian medical university union hospital from April 1, 2012, to May 30, 2022.
- External validation cohort: Patients (n=211) who accepted neoadjuvant systemic therapy followed surgery were from Fujian Cancer Hospital, Zhangzhou Affiliated Hospital of Fujian Medical University and No. 900 Hospital of The Joint Logistic Support Force from April 1, 2012, to May 30, 2022.
- Test cohort: Patients (n=119) who accepted sentinel lymph node biopsy followed axillary lymph node dissection after neoadjuvant systemic therapy was retrospectively collected from June 1,2022 to May 31, 2023.
  Interventions: Procedure: Test cohort

INTERVENTIONS:
Procedure: Test cohort
  Groups: Test cohort

SUMMARY:
The aim of the study was to develop and validate a nomogram to assess axillary pathological complete response (pCR) in patients with initially lymph node-positive, human epidermal growth factor receptor 2 (HER2)-positive breast cancer and test its performance in guiding patient selection for sentinel lymph node biopsy (SLNB) following neoadjuvant systemic therapy (NST).

DETAILED DESCRIPTION:
We retrospectively reviewed the medical records of patients from Fujian Medical University Union Hospital (n = 386) as the training cohort and those from Fujian Cancer Hospital, Zhangzhou Affiliated Hospital of Fujian Medical University, and No. 900 Hospital of The Joint Logistic Support Force (n = 211) as an external validation cohort from April 1, 2012, to March 31, 2022. Additionally, 119 patients were enrolled as the test cohort to assess the predictive power of the model from May 1, 2022, to May 31, 2023.The inclusion criteria included: 1) histologically proven primary breast cancer without distant metastatic lesions, 2) HER2-positive status (defined as immunohistochemistry (IHC) of 3+ overexpression or 2+ expression, and a ratio of ≥ 2.0 by fluorescence in situ hybridization), 3) initial axillary lymph node-positive status confirmed using core- or fine-needle biopsy before NST, 4) a full course of standard neoadjuvant therapy before surgery, and 5) complete clinicopathological characteristics and treatment information. The study was approved by ethics committee of Fujian Medical University Union Hospital. All patients in the training and validation cohorts underwent mastectomy, breast-conserving surgery, radiation, and ALND surgery after completing NST. All patients in the additional independent cohort underwent SLNB followed by ALND, which detected at least 2 SLNs using methylene blue dye alone. SLNs were defined as blue-stained lymph nodes guided directly by blue-stained lymphatic vessels. Methylene blue dye was injected alone at peritumoral or subareolar sites 5-15 min before SLNB. After constructing the nomogram for predicting axillary pCR with the independent predictive factors, the investigators quantified the predictive performance of the model using the AUC of the receiver operating characteristic curve. Calibration plots with bootstrapping and the Hosmer-Lemeshow test were used to illustrate the calibration power of the model, with p > 0.05 indicating a good fit.20 The clinical utility of the model in guiding surgical options was evaluated using decision curve analysis by plotting net benefits.21 Internal validation was estimated using the bootstrap method. The investigators validated the nomogram using an external validation cohort from the other institutions. Following the Youden index, the investigators selected an optimal cutoff probability of predicting axillary pCR as a stratification criterion for identifying patients who underwent SLNB surgery after NST. The investigators additionally examined 119 patients who underwent SLNB with ≥ 2 SLNs removed, followed by ALND, as an independent cohort to evaluate the effect of the nomogram on identifying patients accurately. FNRs of SLNB were compared using two different strategies: performing SLNB in all patients without any selection criteria and performing SLNB in patients selected by the nomogram with the cutoff probability of axillary pCR. These results were compared with those of the two previous tests.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven primary breast cancer without distant metastatic lesions,
* HER2-positive status (defined as immunohistochemistry (IHC) of 3+ overexpression or 2+ expression, and a ratio of ≥ 2.0 by fluorescence in situ hybridization),
* initial axillary lymph node-positive status confirmed using core- or fine-needle biopsy before NST,
* a full course of standard neoadjuvant therapy before surgery
* complete clinicopathological characteristics and treatment information.

Exclusion Criteria:

* do not plan or are unable to operate;
* with distant metastasis
* do not accept full cycles or standard neoadjuvant systemic therapy
* loss of clinicopathological characteristics and treatment information.
* with serious cardiopulmonary diseases, uncontrolled infectious diseases and other non-tumor related diseases who could not tolerate comprehensive treatment such as surgery and chemotherapy

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The investigators retrospectively reviewed the medical records of 597 patients at four institutions from April 1, 2012, to May 30, 2022. Patients from institution 1 (n = 386) served as the training cohort, whereas those from the other institutions (n = 211) served as an external validation cohort. A test cohort (n=119) who accepted SLNB followed ALND was collected to assess the predictive power of the model ，from June 1,2022 to We retrospectively reviewed the medical records of patients from Fujian Medical University Union Hospital (n = 386) as the training cohort and those from Fujian Cancer Hospital, Zhangzhou Affiliated Hospital of Fujian Medical University, and No. 900 Hospital of The Joint Logistic Support Force (n = 211) as an external validation cohort from April 1, 2012, to March 31, 2022. Additionally, 119 patients were enrolled as the test cohort to assess the predictive power of the model from May 1, 2022, to May 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Axillary pCR | 10 years
  the percent of patients who achieved axillary pathological complete response after NST.

SECONDARY OUTCOMES:
the False Negative Rate of SLNB | 12 months
  the percent of patients with residual lymph node disease were not identified.

CONTACTS AND LOCATIONS:
Overall Officials: China Fujian, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Chuan Wang, Fuzhou, Fujian, China